CLINICAL TRIAL: NCT04618198
Title: A Randomized Clinical Trial of Early Empiric Anti-Mycobacterium Tuberculosis Therapy for Sepsis in Sub-Saharan Africa
Brief Title: Early Empiric Anti-Mycobacterium Tuberculosis Therapy for Sepsis in Sub-Saharan Africa
Acronym: ATLAS
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Virginia (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Scott Heysell, MD, Associate Professor, Infectious Disease, University of Virginia
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 22611; U01AI150508-01A1 (NIH)
Record Dates: First submitted 2020-10-26; First posted 2020-11-05 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Tuberculosis; HIV I Infection; Sepsis
MeSH Terms: conditions — Tuberculosis; Sepsis

STUDY DESIGN:
Intervention Model Description: This is a phase 3, multi-site, open-label, randomized controlled clinical 2x2 factorial superiority trial of a) immediate initiation of anti-TB therapy and b) sepsis-specific dose anti-TB therapy for people living with HIV and presenting with sepsis to our regional study sites in Tanzania and Uganda.
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Diagnosis dependent / conventional dose anti-TB therapy (No Intervention): Standard care per admitting team including ceftriaxone x 7 days
  If subsequent TB test positive, then WHO recommended weight-based anti-TB therapy x 28 days
- Immediate anti-TB therapy/conventional dose anti-TB therapy (Experimental): Standard care per admitting team including ceftriaxone x 7 days plus immediate empiric WHO recommended weight-based dose anti-TB therapy x 28 days
  Interventions: Other: Immediate anti-TB therapy
- Diagnosis dependent/sepsis specific dose anti-TB therapy (Experimental): Standard care per admitting team including ceftriaxone x 7 days
  If subsequent TB test positive, then sepsis specific dose anti-TB therapy x 28 days
  Interventions: Other: Sepsis-specific dose anti-TB therapy
- Immediate anti-TB therapy/sepsis specific dose anti-TB therapy (Experimental): Standard care per admitting team including ceftriaxone x 7 days plus immediate empiric sepsis specific dose anti-TB therapy x 28 days
  Interventions: Other: Immediate anti-TB therapy; Other: Sepsis-specific dose anti-TB therapy

INTERVENTIONS:
Other: Immediate anti-TB therapy — Study participants will receive immediate empiric anti-TB therapy
  Arms: Immediate anti-TB therapy/conventional dose anti-TB therapy; Immediate anti-TB therapy/sepsis specific dose anti-TB therapy
Other: Sepsis-specific dose anti-TB therapy — Study participants will receive conventional WHO weight-based dose anti-TB therapy
  Arms: Diagnosis dependent/sepsis specific dose anti-TB therapy; Immediate anti-TB therapy/sepsis specific dose anti-TB therapy

SUMMARY:
In sub-Saharan Africa, tuberculosis (TB) is the etiology of 25-50% of bloodstream infections (BSIs) and the leading cause of sepsis among people living with HIV. TB BSI is associated with 20-50% mortality, and 20-25% of deaths occur within five days of admission. TB BSI is difficult to identify clinically and microbiologically. Given that the high prevalence of TB BSI is under-recognized, most patients with sepsis in sub-Saharan Africa do not receive early anti-TB therapy. The hypothesis of this study is that immediate and optimally dosed anti-TB therapy will improve 28 day mortality in patients with sepsis in Uganda and Tanzania. Therefore, the overall goal is to conduct a phase 3 multi-site open label 2x2 factorial clinical trial of 1) empiric immediate initiation of anti-TB therapy plus standard care compared to diagnosis dependent anti-TB therapy plus standard care and 2) sepsis-specific dose anti-TB therapy plus standard care compared to conventional WHO weight-based dose anti-TB therapy plus standard care for the treatment of sepsis in people living with HIV admitted to our longstanding collaborative research sites at either the Mbarara Regional Referral Hospital in Mbarara, Uganda, or Kilimanjaro region hospitals in Moshi, Tanzania.

DETAILED DESCRIPTION:
The primary objective of this clinical trial is to:

1) To conduct a randomized 2x2 factorial clinical trial of 1) empiric immediate initiation of anti-TB therapy plus standard care vs diagnosis dependent anti-TB therapy plus standard care, 2) sepsis-specific anti-TB therapy plus standard care vs conventional WHO weight-based anti-TB therapy plus standard care for patients presenting with sepsis in Uganda and Tanzania.

1a) To determine if empiric immediate initiation of anti-TB therapy plus standard care improves 28 day mortality compared to diagnosis dependent anti-TB therapy plus standard care.

1b) To determine if sepsis-specific dose anti-TB therapy plus standard care improves 28 day mortality compared to conventional WHO weight-based anti-TB therapy plus standard care.

The secondary objectives include:

1. To determine if empiric immediate initiation of anti-TB therapy plus standard care improves in-hospital mortality compared to diagnosis dependent anti-TB therapy plus standard care.
2. To determine if sepsis-specific dose anti-TB therapy plus standard care improves in-hospital mortality compared to conventional WHO weight-based anti-TB therapy plus standard care.
3. To determine if empiric immediate initiation of anti-TB therapy plus standard care improves 6 month mortality compared to diagnosis dependent anti-TB therapy plus standard care.
4. To determine if sepsis-specific dose anti-TB therapy plus standard care improves 6 month mortality compared to conventional WHO weight-based anti-TB therapy plus standard care.
5. To determine the safety of increased dose sepsis-specific anti-TB therapy for patients with sepsis
6. To determine if early achievement of target serum drug concentrations of isoniazid and rifampin, measured at day-2 of TB treatment, associates with more rapid clinical improvement among patients with confirmed TB.

Participants will be men or women aged ≥18 years living with HIV in Tanzania or Uganda who are admitted to one of the study hospitals with sepsis, defined by a clinical concern for infection, a modified quick sepsis-related organ failure assessment (qSOFA) score ≥2 (Glasgow Coma Scale score <15, a respiratory rate ≥22, or a systolic blood pressure ≤90 mmHg or a mean arterial pressure of ≤65 mmHg). This is a multi-site trial at Kilimanjaro region hospitals in Tanzania (Kibong'oto Infectious Diseases Hospital and Kilimanjaro Christian Medical Centre) and Mbarara Regional Referral Hospital in Mbarara, Uganda. At both regional study sites, clinical trial infrastructure has been developed over multiple TB and non-TB related interventional studies supported by the NIH and other funders including EDCTP, WHO, MRC, and BMGF with associated regulatory standards. Furthermore, both regional hospital systems have large recruitment populations serving mid-sized cities where patients receive local care and as referral hospitals for those from more peripheral settings. The study population will be enrolled from the Emergency or inpatient wards. Admission numbers of eligible patients presenting with sepsis at each site allow for a conservative estimates of 100 patients per country per year to be well within attainment.

After enrollment, patients will be randomized to 1) empiric immediate initiation of anti-TB therapy plus standard care vs diagnosis dependent anti-TB therapy plus standard care and 2) conventional WHO recommended weight-based dose anti-TB therapy with rifampin, isoniazid, pyrazinamide, and ethambutol plus pyridoxine, plus standard therapy; or sepsis-specific dose anti-TB therapy with rifampin (~30mg/kg), isoniazid (~7.5mg/kg), pyrazinamide, and ethambutol plus pyridoxine, plus standard care.

Each individual participant will complete all participant follow-up at 6 months from enrollment.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Male or female aged ≥18 years living with HIV
4. Admitted to hospital with 1) clinical concern for infection; 2) ≥2 qSOFA score criteria (Glasgow Coma Scale score <15, a respiratory rate ≥22, or a systolic blood pressure ≤90 mmHg or a mean arterial pressure of ≤65 mmHg)
5. Resident within a pre-defined geographic area to ensure TB clinic follow-up
6. For females of reproductive potential: use of highly effective contraception through 28 days

Exclusion Criteria:

1. Known active TB or receiving anti-TB therapy
2. Pregnancy or lactation. Women will undergo urine pregnancy screening. Pregnant women will be excluded due to the possible toxicity and teratogenicity of high dose rifampin and isoniazid included in anti-TB therapy as well as possible teratogenicity of dolutegravir which is recommended as first-line antiretroviral therapy in this study.
3. Known allergic reactions to the components of the anti-TB therapy
4. Treatment with another investigational drug or other intervention within one month
5. Known liver disease
6. Alcohol use > 14 standardized drinks per week and/or > 4 drinks per day for men and >7 standardized drinks per week and/or >3 drinks per day for women, defined as 14 grams of ethanol, as found in example 5 ounces of wine, 12 ounces of beer, or 1.5 ounces of 80 proof spirits
7. Positive serum cryptococcal antigen test
8. Current treatment with a drug known to have significant interaction with anti-TB therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 436 (Estimated)
Dates: Start 2021-12-10 (Actual); Primary Completion 2025-03-25 (Estimated); Study Completion 2025-06-25 (Estimated)

PRIMARY OUTCOMES:
28-day mortality | 28 days from enrollment
  number of participants with mortality

SECONDARY OUTCOMES:
In-hospital mortality | 28 days from enrollment
  number of participants with mortality while admitted to the hospital
6-month mortality | 6 months from enrollment
  number of participants with mortality
Time to death | 6 months from enrollment
  time from enrollment to date of mortality
Duration of hospitalization | 6 months from enrollment
  time from enrollment to date of discharge from hospital
Time to anti-TB therapy | 28 days from enrollment
  Time to administration of anti-TB therapy
Adverse events | 28 days from enrollment
  Number of adverse events per participant associated with anti-TB therapy
Sepsis etiology | baseline specimen collection
  pathogen identified in blood by molecular TAC platform
Time to ambulation | 28 days from enrollment
  time from enrollment to date of first ambulation
Time to temperature normalization | 28 days from enrollment
  Time until participant has a normal temperature (above 36C and below 38C)
Karnofsky score | 28 days from enrollment
  Karnofsky score at discharge or death, scale 0 (worst) to 100 (best)
Peak drug concentration isoniazid | 2 days from enrollment
  Serum isoniazid peak concentration (Cmax)
Peak drug concentration rifampin | 2 days from enrollment
  Serum rifampin peak concentration (Cmax)
Total drug exposure isoniazid | 2 days from enrollment
  Serum isoniazid total area under the concentration time curve (AUC)
Total drug exposure rifampin | 2 days from enrollment
  Serum total area under the concentration time curve (AUC)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Moore, MD, Principal Investigator — University of Virginia
Locations (2):
- Kibong'oto Infectious Diseases Hospital, Sanya Juu, Tanzania
- Mbarara University Science Technology, Mbarara, Uganda

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol
Time Frame: Within 1 year from study conclusion
Access Criteria: Reasonable request to the PIs

REFERENCES:
- [Background] Moore CC, Jacob ST, Banura P, Zhang J, Stroup S, Boulware DR, Scheld WM, Houpt ER, Liu J. Etiology of Sepsis in Uganda Using a Quantitative Polymerase Chain Reaction-based TaqMan Array Card. Clin Infect Dis. 2019 Jan 7;68(2):266-272. doi: 10.1093/cid/ciy472. PMID 29868873
- [Background] Hazard RH, Kagina P, Kitayimbwa R, Male K, McShane M, Mubiru D, Welikhe E, Moore CC, Abdallah A. Effect of Empiric Anti-Mycobacterium tuberculosis Therapy on Survival Among Human Immunodeficiency Virus-Infected Adults Admitted With Sepsis to a Regional Referral Hospital in Uganda. Open Forum Infect Dis. 2019 Mar 14;6(4):ofz140. doi: 10.1093/ofid/ofz140. eCollection 2019 Apr. PMID 31024977
- [Background] Mpagama SG, Ndusilo N, Stroup S, Kumburu H, Peloquin CA, Gratz J, Houpt ER, Kibiki GS, Heysell SK. Plasma drug activity in patients on treatment for multidrug-resistant tuberculosis. Antimicrob Agents Chemother. 2014;58(2):782-8. doi: 10.1128/AAC.01549-13. Epub 2013 Nov 18. PMID 24247125
- [Background] Heysell SK, Mtabho C, Mpagama S, Mwaigwisya S, Pholwat S, Ndusilo N, Gratz J, Aarnoutse RE, Kibiki GS, Houpt ER. Plasma drug activity assay for treatment optimization in tuberculosis patients. Antimicrob Agents Chemother. 2011 Dec;55(12):5819-25. doi: 10.1128/AAC.05561-11. Epub 2011 Oct 3. PMID 21968363
- [Background] Byashalira K, Mbelele P, Semvua H, Chilongola J, Semvua S, Liyoyo A, Mmbaga B, Mfinanga S, Moore C, Heysell S, Mpagama S. Clinical outcomes of new algorithm for diagnosis and treatment of Tuberculosis sepsis in HIV patients. Int J Mycobacteriol. 2019 Oct-Dec;8(4):313-319. doi: 10.4103/ijmy.ijmy_135_19. PMID 31793499
- [Derived] Heysell SK, Mpagama SG, Nuwagira E, Said B, Conaway M, Null M, Thomas TA, Boulware DR, Otoupalova E, Arinaitwe R, Mushagara R, Edwards L, Buzaare P, Ngoma AM, Muganzi D, Gidoi G, Jjunju S, Gulinja A, Rimoy AG, Mwita FC, Kidola J, Atwiine O, Ocaaki D, Munyambalu DK, Liu J, Ampaire L, Mujaga B, Rao P, Liyoyo A, Sariko M, Muzoora C, Moore CC. Immediate or high-dose antituberculosis therapy for HIV-related sepsis in Tanzania and Uganda (ATLAS): a phase 3, open-label, randomised, controlled, 2 x 2 factorial, superiority trial. Lancet Infect Dis. 2026 Jan 28:S1473-3099(25)00747-9. doi: 10.1016/S1473-3099(25)00747-9. Online ahead of print. PMID 41619753
- [Derived] Said B, Nuwagira E, Liyoyo A, Arinaitwe R, Gitige C, Mushagara R, Buzaare P, Chongolo A, Jjunju S, Twesigye P, Boulware DR, Conaway M, Null M, Thomas TA, Heysell SK, Moore CC, Muzoora C, Mpagama SG. Early empiric anti-Mycobacterium tuberculosis therapy for sepsis in sub-Saharan Africa: a protocol of a randomised clinical trial. BMJ Open. 2022 Jun 6;12(6):e061953. doi: 10.1136/bmjopen-2022-061953. PMID 35667721